CLINICAL TRIAL: NCT06492382
Title: The Effects of Home Monitors Used with Home Oxygen Therapy: a Randomized Control Trial
Brief Title: The Effects of Home Monitors Used with Home Oxygen Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Per PI, the team couldn't get the home oxygen monitors needed for the study
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Dawn Walstrom Novak, Associate Professor of Pediatrics, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-105:Home Oxygen Monitors
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Frequency of Adverse Events, Health Care Utilization, Infant Growth, Parental Quality of Life, and Altitude of the Participant's Home
Keywords: Home oxygen monitors
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home oxygen monitor (Experimental): Infant will be on a home oxygen weaning guideline for their pediatrician to used based on information form the home oxygen monitor
  Interventions: Diagnostic Test: Home Oxygen Monitors
- No Home oxygen monitor (Active Comparator): Infant will have a home oxygen weaning guideline for their pediatrician to use based on parameters other than a home oxygen monitor
  Interventions: Diagnostic Test: Home Oxygen Monitors

INTERVENTIONS:
Diagnostic Test: Home Oxygen Monitors — Weaning of home oxygen using information gathered from home moniotr devise

SUMMARY:
This study's purpose is to determine the effects of using monitors with home oxygen therapy (HOT). This trial will test the hypothesis that infants discharged from the neonatal intensive care unit (NICU) with HOT will have a shorter treatment duration if used in conjunction with monitors.

DETAILED DESCRIPTION:
This will be a randomized control trial in which infants being discharged from the neonatal intensive care unit with home oxygen therapy will be placed in one of two groups. Those randomized into the treatment group will be sent home with a monitor to be used continuously during their need for supplemental oxygen. The control group will consist of infants randomized to receive the current standard of care, which is discharge with home oxygen and NO home monitor. The research team will contact the families of the subjects at one-month intervals to collect pertinent data.

Aim 1: Subjects will be randomly assigned to a control group (no home monitors, which is current clinical practice) and an experimental group (home monitors). The investigators will compare the duration of treatment with HOT between groups.

Aim 2: Obtain additional data from study participants to better understand the impact of home monitoring. This data includes frequency of adverse events (defined later in the protocol) including health care utilization, as well as parental quality of life, and altitude of the participant's home.

Exploratory Aim 1: Determine the perceptions of families regarding home monitor use.

ELIGIBILITY:
Inclusion Criteria:

* • Infants being discharged with home oxygen therapy.

  * Infants born at other institutions and then transferred to UNMH will be eligible if discharged home with home oxygen therapy.
  * Infants born at gestational age 28 0/7 weeks or greater.
  * Infants of employees of the UNMH will be allowed to participate in the study but will not be targeted. All efforts will be made to ensure that no coercion or undue influence will be used in recruiting this population.

Exclusion Criteria:

* • Infants diagnosed with conditions that will predispose them to prolonged hypoxemia; examples include cardiac anomaly, anatomic anomalies affecting the airway, tracheostomy dependency, cystic fibrosis, and trisomy 21.

  * Infants discharged with hospice care / palliative services.
  * Infants discharged greater than 6 months after they were born.
  * Parents less than 18 years old or prisoners.
  * Parents who are unable to provide consent due to having a legal representative.
  * Infants who are in foster care and/or are wards of the state.
  * Families not fluent in English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-08 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Oxygen Wean | 1 -2 months
  Length of time it takes infant to get off home oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Novak, MD, Principal Investigator — University of New Mexico Children's Hospital

IPD SHARING:
Plan to Share IPD: No